CLINICAL TRIAL: NCT01623752
Title: A PROSPECTIVE EVALUATION OF THE RADIOGRAPHIC EFFICACY OF ETANERCEPT IN PATIENTS WITH RHEUMATOID ARTHRITIS OR PSORIATIC ARTHRITIS.
Brief Title: Prospective Evaluation of the Radiographic Efficacy of Enbrel
Acronym: PRERA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801317
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Results first posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-07

CONDITIONS: Rheumatoid Arthritis; Psoriasis Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Rheumatoid Arthritis
  Interventions: Drug: Etanercept
- Patients with Psoriasis Arthritis
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — The patients will be treated in accordance with the requirements of the labelling of Enbrel® in Germany. The dosage and duration of therapy is to be determined by the physician to meet the patients' individual needs for treatment.
  Other Names: Enbrel
  Groups: Patients with Rheumatoid Arthritis
Drug: Etanercept — The patients will be treated in accordance with the requirements of the labelling of Enbrel® in Germany. The dosage and duration of therapy is to be determined by the physician to meet the patients' individual needs for treatment.
  Other Names: Enbrel
  Groups: Patients with Psoriasis Arthritis

SUMMARY:
It is known from the COMET-trial that patients who start Enbrel treatment early have a great chance of reaching clinical remission and radiographic nonprogression. It is still unclear, however, how many patients with early arthritis achieve remission and radiographic nonprogression under the conditions of routine rheumatologic care and the local recommendations of Enbrel treatment (pre-treatment of at least 2 DMARDs, one of them MTX).

Therefore, no robust x-ray data are available to show/demonstrate

* the average extent of x-ray damage in routine patients on Enbrel outside clinical studies.
* if the outstanding effect on structural damage of Enbrel can be reproduced in routine practice.
* that the 'Silent Progressor' is an issue relevant not only in clinical trials, but also for day-to-day decision making.
* the optimal onset of Enbrel treatment in the course of the disease to prevent radiographic damage

DETAILED DESCRIPTION:
Non-interventional study: subjects to be selected according to the usual clinical practice of their physician

ELIGIBILITY:
Inclusion Criteria:

* Subject eligibility should be reviewed and documented by an appropriately qualified member of the investigator's study team before subjects are included in the study.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study is a requirement for inclusion into this study.

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Definitive diagnosis of RA or PsA.
* Eligible for Etanercept treatment according to Summary of Product Characteristics (SmPC).
* Inclusion of subjects pretreated with other biologics other than Etanercept is possible
* One plain radiograph of hands and feet (Anteroposterior) within 3 month prior to initiation of treatment with Etanercept and one planned consecutive radiograph of hand and feet taken over 12 to 18 months according to German recommendations for patients treated with biologics.

Exclusion Criteria:

* Receipt of any investigational drug within 3 months of study inclusion.
* Exclusion Criteria according to the Enbrel® SmPC, with particular attention to:
* Hypersensitivity to the active substance (etanercept) or to any of the excipients.
* Sepsis or risk of sepsis.
* Active infections, including chronic or localised infections.
* Subjects who have received any previous treatment with etanercept
* Subjects who are investigational site staff members or subjects who are Pfizer employees directly involved in the conduct of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients for whom the decision has already been made to initiate treatment with Enbrel® can be enrolled in this observational trial. These patients must have a proven diagnosis of Rheumatoid Arthritis or Psoriasis Arthritis
Sampling Method: Non-Probability Sample
Enrollment: 1821 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wassenberg S, Rau R, Klopsch T, Plenske A, Jobst J, Klaus P, Meng T, Loschmann PA. Etanercept is Effective and Halts Radiographic Progression in Rheumatoid Arthritis and Psoriatic Arthritis: Final Results from a German Non-interventional Study (PRERA). Rheumatol Ther. 2023 Feb;10(1):117-133. doi: 10.1007/s40744-022-00491-4. Epub 2022 Oct 17. PMID 36251174
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801317&StudyName=Prospective%20Evaluation%20of%20the%20Radiographic%20Efficacy%20of%20Enbrel%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants those who were recruited despite of an unknown or unclear disease diagnosis, were only included in safety analysis for the study, not for efficacy evaluation.
Groups:
- Participants With Rheumatoid Arthritis: Participants with rheumatoid arthritis, who were on Etanercept routine treatment (as per the requirements of the labelling of Enbrel in Germany; dosage and duration of therapy was determined by the physician to meet the participants' individual needs for treatment), were observed for safety and radiological efficacy up to Week 156. During Phase 1 participants were followed up after every 13 weeks up to Week 78 and during Phase 2 participants were followed up after every 16 weeks from Week 78 till Week 156.
- Participants With Psoriatic Arthritis: Participants with psoriatic arthritis, who were on Etanercept routine treatment (as per the requirements of the labelling of Enbrel in Germany; dosage and duration of therapy was determined by the physician to meet the participants' individual needs for treatment), were observed for safety and radiological efficacy up to Week 156. During Phase 1 participants were followed up after every 13 weeks up to Week 78 and during Phase 2 participants were followed up after every 16 weeks from Week 78 till Week 156.
- Participants With Unclear Diagnosis: Participants with unclear diagnosis, who were on Etanercept routine treatment (as per the requirements of the labelling of Enbrel in Germany; dosage and duration of therapy was determined by the physician to meet the participants' individual needs for treatment), were observed for safety and radiological efficacy up to Week 156. During Phase 1 participants were followed up after every 13 weeks up to Week 78 and during Phase 2 participants were followed up after every 16 weeks from Week 78 till Week 156.
Period: Phase 1 (78 Weeks)
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Unclear Diagnosis
Started | 1378 | 440 | 3
Completed | 747 | 233 | 1
Not Completed | 631 | 207 | 2
Not completed — No Data | 249 | 66 | 2
Not completed — Other | 33 | 20 | 0
Not completed — Adverse Event | 122 | 39 | 0
Not completed — Lack of Efficacy | 227 | 82 | 0
Period: Phase 2 (78 Weeks)
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Unclear Diagnosis
Started | 291 (Participants only who consented to continue in Period 2.) | 116 (Participants only who consented to continue in Period 2.) | 0 (Participants only who consented to continue in Period 2.)
Completed | 225 | 98 | 0
Not Completed | 66 | 18 | 0
Not completed — Lack of Efficacy | 14 | 2 | 0
Not completed — Other | 5 | 1 | 0
Not completed — No Data | 43 | 11 | 0
Not completed — Adverse Event | 4 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of Etanercept.
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Unclear Diagnosis | Total
Number analyzed (Participants) | 1378 | 440 | 3 | 1821
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 1 | 0 | 0 | 1
  18 to 64 years | 976 | 387 | 2 | 1365
  65 years or more | 395 | 49 | 0 | 444
  No data | 6 | 4 | 1 | 11
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 1062 | 259 | 2 | 1323
  Male | 316 | 181 | 0 | 497
  No Data | 0 | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Van Der Heijde Total Modified Total Sharp Score (mTSS) or Adapted mTSS at End of Phase 1 (Week 78): Efficacy Analysis Set (EAS)
Description: To assess radiological damage mTSS score was used in participants with rheumatoid arthritis and mTSS adapted score was used in participants with psoriatic arthritis. Radiographs of the hands and feet were assessed by central raters. Total mTSS score range was 0 (no radiological damage) to 448 (extreme radiological damage); and total mTSS adapted score range was 0 (no radiological damage) to 528 (extreme radiological damage), where higher mTSS and mTSS adapted scores indicate a worse health status in participants with rheumatoid arthritis and participants with psoriatic arthritis, respectively.
Time Frame: Baseline, Week 78
Population: Efficacy analysis set for Phase 1= all participants who had received at least 1 dose of Etanercept and had baseline X-ray (Rx1) and end of phase 1 X-ray (Rx2). Here, "Overall Number of Participants Analyzed" =number of participants evaluable for this outcome measure; "Number Analyzed"=number of participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 504 | 166
Units on a scale
  Baseline | 25.1 (42.4) | 14.7 (25.7)
  Change at Week 78: number analyzed (Participants) | 489 | 160
  Change at Week 78 | 0.6 (7.2) | -0.4 (5.9)

2. Primary Outcome: Change From Baseline in Van Der Heijde Total Modified Total Sharp Score or Adapted mTSS at End of Phase 1 (Week 78): Completer Analysis Set (CAS)
Description: To assess radiological damage, mTSS score was used in participants with rheumatoid arthritis and mTSS adapted score was used in participants with psoriatic arthritis. Radiographs of the hands and feet were assessed by central raters. Total mTSS score range was 0 (no radiological damage) to 448 (extreme radiological damage); and total mTSS adapted score range was 0 (no radiological damage) to 528 (extreme radiological damage), where higher mTSS and mTSS adapted scores indicate a worse health status in participants with rheumatoid arthritis and participants with psoriatic arthritis, respectively.
Time Frame: Baseline, Week 78
Population: Completer analysis set for Phase 1: all participants who had received at least 1 dose of Etanercept and had clinical data for Rx1 and Rx2 and provided data for end of Phase 1 of study. "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure. "Number Analyzed"= participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 500 | 164
Units on a scale
  Baseline | 25.3 (42.5) | 14.7 (25.8)
  Change at Week 78: number analyzed (Participants) | 486 | 158
  Change at Week 78 | 0.6 (7.2) | -0.5 (5.8)

3. Primary Outcome: Change From Baseline in Van Der Heijde Total Modified Total Sharp Score or Adapted mTSS at the End of Phase 2 (Week 156): EAS
Description: as for outcome 2
Time Frame: Baseline, Week 156
Population: Efficacy analysis set for Phase 2 included all participants who had received at least 1 dose of Etanercept and had Rx1 and end of Phase 2 X-ray (Rx3). Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 97 | 48
Units on a scale | 1.4 (9.9) | 0.7 (8.2)

4. Primary Outcome: Change From Baseline in Van Der Heijde Total Modified Total Sharp Score or Adapted mTSS at End of Phase 2 (Week 156): CAS
Description: as for outcome 2
Time Frame: Baseline, Week 156
Population: Completer analysis set for Phase 2 included all participants who had received at least 1 dose of Etanercept, and had clinical data for the obligatory X-ray (Rx1) and Rx3, and completed Phase 2 of the study. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 96 | 48
Units on a scale | 1.4 (9.9) | 0.7 (8.2)

5. Primary Outcome: Change From Pre-treatment in Normalized Radiographic Progression of mTSS or Adapted mTSS at End of Phase 1 (Week 78): EAS
Description: The normalized change in total scores (mTSS or mTSS adapted) were computed as normalized per year (normalized progression). The change of normalized progression was classified as: increase (greater than [>] 0.5), no change (-0.5 to 0.5) and decrease (less than [<] -0.5). Participants with no change or a decrease were considered to be in radiographic remission.
Time Frame: Pre-treatment, Week 78
Population: Efficacy analysis set for Phase 1 included all participants who had received at least 1 dose of Etanercept and had Rx1 and Rx2. Here, "Overall Number of Participants Analyzed" = number of participants evaluable for this outcome measure and "Number Analyzed" = number of participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Scores per year
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 189 | 46
Scores per year
  Pre-treatment | 0.959 (4.396) | 1.056 (5.127)
  Change at Week 78: number analyzed (Participants) | 176 | 45
  Change at Week 78 | -0.267 (5.989) | -0.995 (8.628)
Statistical Analysis 1: Comparison: Participants With Rheumatoid Arthritis; P-value was calculated using Paired t-test for the change in normalized progression; Test type: Other; p = 0.278, Paired t-test
Statistical Analysis 2: Comparison: Participants With Psoriatic Arthritis; P-value was calculated using Paired t-test for the change in normalized progression; Test type: Other; p = 0.222, Paired t-test

6. Primary Outcome: Change From Pre-treatment in Normalized Radiographic Progression of mTSS or Adapted mTSS at End of Phase 1 (Week 78): CAS
Description: The normalized change in total scores (mTSS or mTSS adapted) were computed as normalized per year (normalized progression). The change of normalized progression was classified as: increase (>0.5), no change (-0.5 to 0.5) and decrease (<-0.5). Participants with no change or a decrease were considered to be in radiographic remission.
Time Frame: Pre-treatment, Week 78
Population: CAS for phase 1 included all participants who had received at least 1 dose of Etanercept, and had Rx1 and Rx2, and provided data for end of Phase 1 of study. Here, "Overall Number of Participants Analyzed"=number of participants evaluable for this outcome measure and "Number Analyzed"=number of participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Scores per year
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 187 | 45
Scores per year
  Pre-treatment | 0.981 (4.413) | 1.080 (5.182)
  Change at Week 78: number analyzed (Participants) | 174 | 44
  Change at Week 78 | -0.306 (6.002) | -1.033 (8.724)
Statistical Analysis 1: Comparison: Participants With Rheumatoid Arthritis; P-value was calculated using Paired t-test for the change in normalized progression; Test type: Other; p = 0.251, Paired t-test
Statistical Analysis 2: Comparison: Participants With Psoriatic Arthritis; P-value was calculated using Paired t-test for the change in normalized progression; Test type: Other; p = 0.218, Paired t-test

7. Primary Outcome: Change From Pre-treatment in Normalized Radiographic Progression of mTSS or Adapted mTSS at End of Phase 2 (Week 156): EAS
Description: as for outcome 6
Time Frame: Pre-treatment, Week 156
Population: Efficacy analysis set for Phase 2 included all participants who had received at least 1 dose of Etanercept and had Rx1 and Rx3. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores per year
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 40 | 15
Scores per year | -0.473 (5.940) | -0.348 (3.985)

8. Primary Outcome: Change From Pre-treatment in Normalized Radiographic Progression of mTSS or Adapted mTSS at the End of Phase 2 (Week 156): CAS
Description: as for outcome 6
Time Frame: Pre-treatment, Week 156
Population: CAS for phase 2 included all participants who had received at least 1 dose of Etanercept, and had Rx1 and Rx2, and completed phase 2 of the study. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores per year
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 40 | 15
Scores per year | -0.473 (5.940) | -0.348 (3.985)

9. Secondary Outcome: Linear Relationship Between Normalized Radiographic Progression and Disease Duration
Description: Linear relationship between radiographic progression and disease duration was evaluated using a linear regression model. Dependent variable was normalized progression under treatment with Etanercept and independent variable was disease duration.
Time Frame: Baseline up to Week 78
Population: Efficacy analysis set for Phase 1 included participants who received at least 1 dose of Etanercept and had Rx1 and Rx2. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: Regression coefficient
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 466 | 157
Regression coefficient | -0.012 | -0.050
Statistical Analysis 1: Comparison: Participants With Rheumatoid Arthritis; Test type: Other; p = 0.675, Regression, Linear
Statistical Analysis 2: Comparison: Participants With Psoriatic Arthritis; Test type: Other; p = 0.357, Regression, Linear

10. Secondary Outcome: Effect on Normalized Radiographic Progression With Respect to Baseline Positivity of Anti-citrullinated Protein Antibody (ACPA) - Rheumatoid Factor (RF)
Description: Effect on normalized radiographic progression with respect to ACPA-RF was evaluated using an analysis of variance (ANOVA) model. Dependent variable was normalized progression under treatment with Etanercept and independent variable was groups of positive testing of ACPA and RF at baseline.
Time Frame: Baseline up to Week 78
Population: Efficacy analysis set for Phase 1 included participants who received at least 1 dose of Etanercept and had Rx1 and Rx2. Here, "Overall Number of Participants Analyzed" = number of participants evaluable for this outcome measure and "Number Analyzed" = number of participants evaluable for the specified rows.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores per year
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 387 | 87
Scores per year
  ACPA and RF negative: number analyzed (Participants) | 98 | 78
  ACPA and RF negative | 1.326 [0.292 to 2.359] | -1.142 [-2.486 to 0.202]
  ACPA or RF positive: number analyzed (Participants) | 104 | 6
  ACPA or RF positive | 1.075 [0.072 to 2.078] | 2.448 [-2.398 to 7.294]
  ACPA and RF positive: number analyzed (Participants) | 185 | 3
  ACPA and RF positive | 0.087 [-0.665 to 0.839] | 3.370 [-3.484 to 10.224]
Statistical Analysis 1: Comparison: Participants With Rheumatoid Arthritis; Statistical analysis (P value) composite for all categories; Test type: Other; p = 0.106, ANOVA
Statistical Analysis 2: Comparison: Participants With Psoriatic Arthritis; Statistical analysis (P value) composite for all categories; Test type: Other; p = 0.181, ANOVA

11. Secondary Outcome: Effect on Normalized Radiographic Progression With Respect to Baseline Usage of Concomitant Medication
Description: Effect on normalized radiographic progression with respect to use of concomitant medication at baseline was evaluated using an ANOVA model. Dependent variable was normalized progression under treatment with Etanercept and independent variable was groups of concomitant medication as found among the medication given concomitantly during study that is recorded at baseline.
Time Frame: Baseline up to Week 78
Population: as for outcome 10
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores per year
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 471 | 157
Scores per year
  Concomitant Medication at baseline: Yes: number analyzed (Participants) | 411 | 94
  Concomitant Medication at baseline: Yes | 0.749 [0.253 to 1.245] | -0.339 [-1.339 to 0.661]
  Concomitant Medication at baseline: No: number analyzed (Participants) | 60 | 63
  Concomitant Medication at baseline: No | -0.978 [-2.276 to 0.320] | -0.370 [-1.592 to 0.851]
Statistical Analysis 1: Comparison: Participants With Rheumatoid Arthritis; Statistical analysis (P value) composite for all categories; Test type: Other; p = 0.015, ANOVA
Statistical Analysis 2: Comparison: Participants With Psoriatic Arthritis; Statistical analysis (P value) composite for all categories; Test type: Other; p = 0.969, ANOVA

12. Secondary Outcome: Effect on Normalized Radiographic Progression With Respect to Previous Treatment With Biologics
Description: Effect on normalized radiographic progression of previous treatment with biologics was evaluated using an ANOVA model. Dependent variable was normalized progression under treatment with Etanercept and independent variable was previous treatment with biologics.
Time Frame: Baseline up to Week 78
Population: as for outcome 10
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores per year
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 471 | 157
Scores per year
  Previous treatment with biologics: number analyzed (Participants) | 112 | 35
  Previous treatment with biologics | 0.235 [-0.720 to 1.191] | -0.986 [-2.621 to 0.649]
  No previous treatment with biologics: number analyzed (Participants) | 359 | 122
  No previous treatment with biologics | 0.621 [0.087 to 1.155] | -0.170 [-1.045 to 0.706]
Statistical Analysis 1: Comparison: Participants With Rheumatoid Arthritis; Statistical analysis (P value) composite for all categories; Test type: Other; p = 0.489, ANOVA
Statistical Analysis 2: Comparison: Participants With Psoriatic Arthritis; Statistical analysis (P value) composite for all categories; Test type: Other; p = 0.386, ANOVA

13. Secondary Outcome: Effect on Normalized Radiographic Progression With Respect to Baseline Disease Activity Score-28 (DAS-28)
Description: Effect on radiographic progression with respect to baseline DAS-28 was evaluated using ANOVA model. Dependent variable was normalized progression under treatment with Etanercept and independent variable was baseline DAS-28. Baseline DAS-28 is less than or equal to (<=) 5.1 or >5.1. DAS28: score range from 0 (none) to 9.4 (extreme disease activity); low =2.6 to 3.2, moderate =3.2 to 5.1, and high disease activity >5.1. DAS28 score of <2.6 indicates disease remission.
Time Frame: Baseline up to Week 78
Population: as for outcome 10
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores per year
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 367 | 126
Scores per year
  Baseline DAS-28 <= 5.1: number analyzed (Participants) | 244 | 99
  Baseline DAS-28 <= 5.1 | 0.716 [0.033 to 1.399] | -0.314 [-1.242 to 0.613]
  Baseline DAS-28 > 5.1: number analyzed (Participants) | 123 | 27
  Baseline DAS-28 > 5.1 | 0.170 [-0.792 to 1.133] | -0.507 [-2.283 to 1.268]
Statistical Analysis 1: Comparison: Participants With Rheumatoid Arthritis; Statistical analysis (P value) composite for all categories; Test type: Other; p = 0.364, ANOVA
Statistical Analysis 2: Comparison: Participants With Psoriatic Arthritis; Statistical analysis (P value) composite for all categories; Test type: Other; p = 0.849, ANOVA

14. Secondary Outcome: Change From Baseline in Total Erosion Score at End of Phase 1 (Week 78) and Phase 2 (Week 156)
Description: Total erosion score as per van der Hejde method consisted of 2 dimensions: a) hands (32 erosion locations, each location graded from 0 [no erosion] to 5 [maximum severity], sum of grading of each location resulted in score of 0 to 160); and b) feet (12 erosion locations, each location graded from 0 [no erosion] to 10 [maximum severity], sum of grading of each location resulted in score of 0 to 120). Sum of erosion scores of hand (0 to 160) and feet (0 to 120) gave a total erosion score as 0 to 280, where 0 was no erosion at all and 280 was worst possible condition, higher scores indicated severe joint destruction.
Time Frame: Baseline, Week 78, 156
Population: Efficacy analysis set included participants who received at least 1 dose of Etanercept and had Rx1 and Rx2 or had Rx1 and Rx3. Here, "Overall Number of Participants Analyzed" = number of participants evaluable for this outcome measure and "Number Analyzed" = number of participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 505 | 166
Units on a scale
  Baseline | 11.1 (23.8) | 4.6 (11.9)
  Change at Week 78: number analyzed (Participants) | 490 | 160
  Change at Week 78 | -0.1 (4.1) | -0.3 (3.1)
  Change at Week 156: number analyzed (Participants) | 97 | 48
  Change at Week 156 | 0.0 (5.7) | 0.2 (6.5)

15. Secondary Outcome: Change From Baseline in Total Joint Space Narrow Score at End of Phase 1 (Week 78) and Phase 2 (Week 156)
Description: Total joint space narrow score as per van der Hejde method consisted of 2 dimensions: a) hands (30 joint space locations, each location graded from 0 [normal joint space] to 4 [bony ankylosis], sum of grading of each location resulted in score of 0 to 120); and b) feet (12 erosion locations, each location graded from 0 [no erosion] to 4 [bony ankylosis], sum of grading of each location resulted in score of 0 to 48). Sum of joint space narrow scores of hand (0 to 120) and feet (0 to 48) gave a total joint space narrow score as 0 to 168, where 0 was normal joint space and 168 was maximum narrowing in joints, higher scores indicated severe joint destruction.
Time Frame: Baseline, Week 78, 156
Population: Efficacy analysis set included participants who received at least 1 dose of Etanercept and had Rx1 and Rx2 or have Rx1 and Rx3. Here, "Overall Number of Participants Analyzed" = number of participants evaluable for this outcome measure and "Number Analyzed" = number of participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 507 | 166
Units on a scale
  Baseline | 14.0 (19.9) | 10.0 (15.0)
  Change at Week 78: number analyzed (Participants) | 492 | 160
  Change at Week 78 | 0.7 (4.3) | -0.1 (3.7)
  Change at Week 156: number analyzed (Participants) | 97 | 48
  Change at Week 156 | 1.4 (5.9) | 0.6 (3.1)

16. Secondary Outcome: Change From Baseline in Hannover Functional Ability Questionnaire (FFbH) at Week 13, 26, 39, 52, 65, 78, 104, 130 and 156
Description: FFbH is a self-administered patient questionnaire composed by 18 questions on functional ability in activities of daily living. Each question was answered by the participant as "Yes, I can perform the activity without difficulty" (score assigned =2), "Yes, but with difficulties" (score assigned =1) and "No or only with external help" (score assigned =0). Final FFbH score (%) was then computed according to formula: (Sum of scores*100) divided by (2*number of valid answers), ranging between 0 (no functional capacity) to 100 (full functional capacity); higher scores indicate better daily activities. FFbH functional remission was defined as FFbH functional capacity of >= 83%.
Time Frame: Baseline, Week 13, 26, 39, 52, 65, 78, 104, 130, 156
Population: Full analysis set included all participants who received at least 1 dose of Etanercept and had at least 1 effectiveness measurement after start of treatment. Here, "Number Analyzed" signifies number of participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1281 | 413
Units on a scale
  Baseline: number analyzed (Participants) | 1271 | 409
  Baseline | 64.99 (22.71) | 68.67 (22.09)
  Change at Week 13: number analyzed (Participants) | 1228 | 397
  Change at Week 13 | 4.38 (12.94) | 3.45 (13.44)
  Change at Week 26: number analyzed (Participants) | 1016 | 340
  Change at Week 26 | 5.63 (15.25) | 3.99 (15.11)
  Change at Week 39: number analyzed (Participants) | 894 | 273
  Change at Week 39 | 6.20 (15.43) | 4.90 (14.46)
  Change at Week 52: number analyzed (Participants) | 807 | 251
  Change at Week 52 | 5.78 (15.27) | 4.43 (16.47)
  Change at Week 65: number analyzed (Participants) | 716 | 220
  Change at Week 65 | 6.15 (15.96) | 4.83 (16.52)
  Change at Week 78: number analyzed (Participants) | 689 | 208
  Change at Week 78 | 6.59 (16.16) | 3.62 (16.37)
  Change at Week 104: number analyzed (Participants) | 276 | 109
  Change at Week 104 | 6.10 (14.98) | 5.09 (14.54)
  Change at Week 130: number analyzed (Participants) | 250 | 106
  Change at Week 130 | 6.22 (15.46) | 4.66 (15.03)
  Change at Week 156: number analyzed (Participants) | 214 | 93
  Change at Week 156 | 5.54 (16.42) | 3.56 (15.78)

17. Secondary Outcome: Change From Baseline in Disease Activity Score-28 (DAS-28) at Week 13, 26, 39, 52, 65, 78, 104, 130 and 156
Description: DAS28 was calculated from swollen joint count and tender joint count using 28 joint count, C-reactive protein (CRP) in milligram per liter (mg/L) and participant global assessment (PtGA) of disease activity measured on a 100 mm visual analog scale (VAS) ranging from 0 (good condition) to 100 (worst condition), where higher scores indicate worse health condition). DAS28 total score range: 0 (no disease activity) to 9.4 (maximum disease activity), higher score indicates more disease activity. DAS-28 score of 2.6 to 3.2= low, 3.2 to 5.1= moderate and >5.1= high disease activity. DAS-28 score of <2.6= disease remission. DAS28-4(CRP) = (0.56*sqrt[TJC28] + 0.28*sqrt[SJC28] + 0.36*ln[CRP+1]) + 0.014*GH + 0.96) and DAS28-4(ESR) = (0.56*sqrt[TJC28] + 0.28*sqrt[SJC28] + 0.70*ln[ESR] + 0.014*GH), where sqrt = square root, ln = natural logarithm.
Time Frame: Baseline, Week 13, 26, 39, 52, 65, 78, 104, 130, 156
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1281 | 431
Units on a scale
  Baseline: number analyzed (Participants) | 1014 | 327
  Baseline | 4.63 (1.24) | 4.18 (1.11)
  Change at Week 13: number analyzed (Participants) | 836 | 269
  Change at Week 13 | -1.26 (1.38) | -1.23 (1.31)
  Change at Week 26: number analyzed (Participants) | 686 | 221
  Change at Week 26 | -1.52 (1.38) | -1.37 (1.28)
  Change at Week 39: number analyzed (Participants) | 591 | 183
  Change at Week 39 | -1.57 (1.41) | -1.52 (1.27)
  Change at Week 52: number analyzed (Participants) | 546 | 184
  Change at Week 52 | -1.64 (1.41) | -1.69 (1.20)
  Change at Week 65: number analyzed (Participants) | 473 | 147
  Change at Week 65 | -1.76 (1.47) | -1.54 (1.26)
  Change at Week 78: number analyzed (Participants) | 449 | 154
  Change at Week 78 | -1.73 (1.38) | -1.62 (1.31)
  Change at Week 104: number analyzed (Participants) | 197 | 77
  Change at Week 104 | -1.94 (1.33) | -1.67 (1.37)
  Change at Week 130: number analyzed (Participants) | 184 | 71
  Change at Week 130 | -1.96 (1.36) | -1.66 (1.27)
  Change at Week 156: number analyzed (Participants) | 149 | 71
  Change at Week 156 | -2.10 (1.42) | -1.54 (1.39)

18. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 13, 26, 39, 52, 65, 78, 104, 130 and 156 in Participants With Rheumatoid Arthritis
Description: CDAI was calculated from tender and swollen joints using 28 joint count, participant global assessment (PtGA) and physician global assessment (PhyGA). PtGA and PhyGA both were assessed on 0-100 mm VAS scale, where higher scores indicated greater affection due to disease activity. CDAI total score ranged from 0 to 76, where higher scores indicated higher disease activity. CDAI score of <=10 indicates low disease activity and a score of <= 2.8 indicates remission.
Time Frame: Baseline, Week 13, 26, 39, 52, 65, 78, 104, 130, 156
Population: Full analysis set: all participants who received at least 1 dose of Etanercept and had at least 1 effectiveness measurement after start of treatment. "Number Analyzed" = number of participants evaluable for the specified time points. Data for this outcome measure was to be collected and evaluated only for participants with rheumatoid arthritis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 1281
Units on a scale
  Baseline: number analyzed (Participants) | 1043
  Baseline | 25.64 (12.14)
  Change at Week 13: number analyzed (Participants) | 963
  Change at Week 13 | -11.51 (12.13)
  Change at Week 26: number analyzed (Participants) | 787
  Change at Week 26 | -13.49 (12.53)
  Change at Week 39: number analyzed (Participants) | 694
  Change at Week 39 | -13.98 (12.78)
  Change at Week 52: number analyzed (Participants) | 623
  Change at Week 52 | -14.32 (12.29)
  Change at Week 65: number analyzed (Participants) | 546
  Change at Week 65 | -15.28 (12.66)
  Change at Week 78: number analyzed (Participants) | 530
  Change at Week 78 | -15.54 (12.28)
  Change at Week 104: number analyzed (Participants) | 208
  Change at Week 104 | -17.53 (11.99)
  Change at Week 130: number analyzed (Participants) | 198
  Change at Week 130 | -17.37 (12.18)
  Change at Week 156: number analyzed (Participants) | 167
  Change at Week 156 | -18.38 (11.99)

19. Secondary Outcome: Change From Baseline in Simple Disease Activity Index (SDAI) at Week 13, 26, 39, 52, 65, 78, 104, 130 and 156 in Participants With Rheumatoid Arthritis
Description: SDAI was calculated from tender and swollen joints using 28 joint count, participant global assessment (PtGA), physician global assessment and (PhyGA) and CRP (in mg/L). PtGA and PhyGA both were assessed on 0-100 mm VAS scale, where higher scores indicated greater affection due to disease activity. SDAI total score ranged from 0 to 86, where higher scores indicated higher disease activity. SDAI score of <=11 indicates low disease activity and a score of <=3.3 indicates remission.
Time Frame: Baseline, Week 13, 26, 39, 52, 65, 78, 104, 130, 156
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 1281
Units on a scale
  Baseline: number analyzed (Participants) | 957
  Baseline | 35.88 (198.26)
  Change at Week 13: number analyzed (Participants) | 751
  Change at Week 13 | -20.62 (225.74)
  Change at Week 26: number analyzed (Participants) | 609
  Change at Week 26 | -26.04 (248.89)
  Change at Week 39: number analyzed (Participants) | 517
  Change at Week 39 | -16.00 (45.07)
  Change at Week 52: number analyzed (Participants) | 481
  Change at Week 52 | -17.70 (47.40)
  Change at Week 65: number analyzed (Participants) | 407
  Change at Week 65 | -18.77 (49.86)
  Change at Week 78: number analyzed (Participants) | 396
  Change at Week 78 | -19.02 (51.83)
  Change at Week 103: number analyzed (Participants) | 175
  Change at Week 103 | -18.08 (15.07)
  Change at Week 130: number analyzed (Participants) | 163
  Change at Week 130 | -17.33 (17.19)
  Change at Week 156: number analyzed (Participants) | 129
  Change at Week 156 | -18.85 (14.06)

20. Secondary Outcome: Percentage of Participants With Rheumatoid Arthritis, With Low Disease Activity Based on Clinical Disease Activity Index (CDAI) and Simple Disease Activity Index (SDAI)
Description: CDAI was calculated from tender and swollen joints using 28 joint count, PtGA and PhyGA. CDAI total score ranged from 0 to 76, where higher scores indicated higher disease activity. CDAI score of <=10 indicates low disease activity and a score of <= 2.8 indicates remission. SDAI was calculated from tender and swollen joints using 28 joint count, PtGA, PhyGA and CRP (in mg/L). SDAI total score ranged from 0 to 86, where higher scores indicated higher disease activity. SDAI score of <=11 indicates low disease activity and a score of <=3.3 indicates remission. PtGA and PhyGA both were assessed on 0-100 mm VAS scale, where higher scores indicated greater affection due to disease activity.
Time Frame: Baseline, Week 13, 26, 39, 52, 65, 78, 104, 130, 156
Population: as for outcome 18
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 1281
Percentage of participants
  Baseline: CDAI: number analyzed (Participants) | 1043
  Baseline: CDAI | 7.0
  Week 13: CDAI: number analyzed (Participants) | 1023
  Week 13: CDAI | 36.1
  Week 26: CDAI: number analyzed (Participants) | 838
  Week 26: CDAI | 41.2
  Week 39: CDAI: number analyzed (Participants) | 744
  Week 39: CDAI | 37.8
  Week 52: CDAI: number analyzed (Participants) | 666
  Week 52: CDAI | 38.0
  Week 65: CDAI: number analyzed (Participants) | 584
  Week 65: CDAI | 43.7
  Week 78: CDAI: number analyzed (Participants) | 566
  Week 78: CDAI | 40.3
  Week 103: CDAI: number analyzed (Participants) | 259
  Week 103: CDAI | 44.4
  Week 130: CDAI: number analyzed (Participants) | 241
  Week 130: CDAI | 41.5
  Week 165: CDAI: number analyzed (Participants) | 207
  Week 165: CDAI | 43.0
  Baseline: SDAI: number analyzed (Participants) | 957
  Baseline: SDAI | 7.0
  Week 13: SDAI: number analyzed (Participants) | 818
  Week 13: SDAI | 35.2
  Week 26: SDAI: number analyzed (Participants) | 662
  Week 26: SDAI | 41.1
  Week 39: SDAI: number analyzed (Participants) | 573
  Week 39: SDAI | 38.7
  Week 52: SDAI: number analyzed (Participants) | 528
  Week 52: SDAI | 39.2
  Week 65: SDAI: number analyzed (Participants) | 445
  Week 65: SDAI | 45.8
  Week 78: SDAI: number analyzed (Participants) | 431
  Week 78: SDAI | 43.2
  Week 103: SDAI: number analyzed (Participants) | 223
  Week 103: SDAI | 43.5
  Week 130: SDAI: number analyzed (Participants) | 207
  Week 130: SDAI | 44.0
  Week 165: SDAI: number analyzed (Participants) | 166
  Week 165: SDAI | 38.0

21. Secondary Outcome: Percentage of Participants With Rheumatoid Arthritis, With Remission Based on Clinical Disease Activity Index (CDAI) and Simple Disease Activity Index (SDAI)
Description: as for outcome 20
Time Frame: Baseline, Week 13, 26, 39, 52, 65, 78, 104, 130, 156
Population: Full analysis set. Here, "Overall Number of Participants Analyzed" = number of participants evaluable for this outcome measure and "Number Analyzed" = number of participants evaluable for the specified time points. Data for this outcome measure was to be collected and evaluated only for participants with rheumatoid arthritis.
Measure: Number; unit: Percentage of participants
Arm/Group | Participants With Rheumatoid Arthritis
Number analyzed (Participants) | 1281
Percentage of participants
  Baseline: CDAI: number analyzed (Participants) | 1043
  Baseline: CDAI | 0.6
  Week 13: CDAI: number analyzed (Participants) | 1023
  Week 13: CDAI | 11.2
  Week 26: CDAI: number analyzed (Participants) | 838
  Week 26: CDAI | 16.0
  Week 39: CDAI: number analyzed (Participants) | 744
  Week 39: CDAI | 19.8
  Week 52: CDAI: number analyzed (Participants) | 666
  Week 52: CDAI | 21.3
  Week 65: CDAI: number analyzed (Participants) | 584
  Week 65: CDAI | 22.8
  Week 78: CDAI: number analyzed (Participants) | 566
  Week 78: CDAI | 25.3
  Week 103: CDAI: number analyzed (Participants) | 259
  Week 103: CDAI | 24.7
  Week 130: CDAI: number analyzed (Participants) | 241
  Week 130: CDAI | 27.0
  Week 165: CDAI: number analyzed (Participants) | 207
  Week 165: CDAI | 31.9
  Baseline: SDAI: number analyzed (Participants) | 957
  Baseline: SDAI | 0.4
  Week 13: SDAI: number analyzed (Participants) | 818
  Week 13: SDAI | 11.1
  Week 26: SDAI: number analyzed (Participants) | 662
  Week 26: SDAI | 13.6
  Week 39: SDAI: number analyzed (Participants) | 573
  Week 39: SDAI | 17.3
  Week 52: SDAI: number analyzed (Participants) | 528
  Week 52: SDAI | 19.3
  Week 65: SDAI: number analyzed (Participants) | 445
  Week 65: SDAI | 19.8
  Week 78: SDAI: number analyzed (Participants) | 431
  Week 78: SDAI | 22.3
  Week 103: SDAI: number analyzed (Participants) | 223
  Week 103: SDAI | 23.3
  Week 130: SDAI: number analyzed (Participants) | 207
  Week 130: SDAI | 25.1
  Week 165: SDAI: number analyzed (Participants) | 166
  Week 165: SDAI | 35.5

22. Secondary Outcome: Change From Baseline in Participant Pain Visual Analogue Scale (VAS) at Week 13, 26, 39, 52, 65, 78, 104, 130 and 156
Description: VAS: participants placed a mark indicating the intensity of their pain on a scale of 0 (no pain) to 100 mm (worst possible pain). Higher scores indicate greater level of pain.
Time Frame: Baseline, Week 13, 26, 39, 52, 65, 78, 104, 130, 156
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1281 | 413
millimeter
  Baseline: number analyzed (Participants) | 1074 | 356
  Baseline | 55.93 (26.26) | 57.69 (25.14)
  Change at Week 13: number analyzed (Participants) | 1011 | 335
  Change at Week 13 | -15.03 (28.50) | -18.20 (27.96)
  Change at Week 26: number analyzed (Participants) | 823 | 287
  Change at Week 26 | -18.56 (29.83) | -19.01 (27.51)
  Change at Week 39: number analyzed (Participants) | 727 | 232
  Change at Week 39 | -18.38 (29.91) | -21.84 (29.62)
  Change at Week 52: number analyzed (Participants) | 648 | 218
  Change at Week 52 | -19.73 (31.02) | -22.24 (30.57)
  Change at Week 65: number analyzed (Participants) | 568 | 190
  Change at Week 65 | -22.83 (30.95) | -22.40 (29.74)
  Change at Week 78: number analyzed (Participants) | 550 | 180
  Change at Week 78 | -22.58 (32.12) | -24.91 (31.69)
  Change at Week 104: number analyzed (Participants) | 222 | 94
  Change at Week 104 | -23.46 (29.01) | -21.09 (32.67)
  Change at Week 130: number analyzed (Participants) | 205 | 87
  Change at Week 130 | -24.67 (28.75) | -21.67 (29.18)
  Change at Week 156: number analyzed (Participants) | 172 | 82
  Change at Week 156 | -26.88 (28.77) | -18.33 (31.13)

23. Secondary Outcome: Change From Baseline in Physician Global Assessment (PhyGA) of Disease Activity at Week 13, 26, 39, 52, 65, 78, 104, 130 and 156
Description: PhyGA: physician marked intensity of participants' pain on a visual analogue scale of 0 (no disease activity) to 100 mm (worst possible condition). Higher scores indicate greater level of disease activity.
Time Frame: Baseline, Week 13, 26, 39, 52, 65, 78, 104, 130, 156
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1281 | 413
millimeter
  Baseline: number analyzed (Participants) | 1100 | 360
  Baseline | 57.28 (19.38) | 55.73 (19.90)
  Change at Week 13: number analyzed (Participants) | 1065 | 350
  Change at Week 13 | -24.49 (22.98) | -24.97 (23.29)
  Change at Week 26: number analyzed (Participants) | 873 | 301
  Change at Week 26 | -29.22 (24.42) | -28.54 (24.28)
  Change at Week 39: number analyzed (Participants) | 775 | 241
  Change at Week 39 | -30.67 (23.92) | -32.06 (24.46)
  Change at Week 52: number analyzed (Participants) | 702 | 220
  Change at Week 52 | -31.78 (24.74) | -34.36 (22.72)
  Change at Week 65: number analyzed (Participants) | 617 | 196
  Change at Week 65 | -34.07 (24.83) | -34.37 (24.02)
  Change at Week 78: number analyzed (Participants) | 603 | 191
  Change at Week 78 | -35.88 (25.29) | -35.87 (23.66)
  Change at Week 104: number analyzed (Participants) | 239 | 98
  Change at Week 104 | -37.10 (23.18) | -34.87 (21.22)
  Change at Week 130: number analyzed (Participants) | 218 | 92
  Change at Week 130 | -37.11 (22.96) | -33.98 (22.19)
  Change at Week 156: number analyzed (Participants) | 186 | 84
  Change at Week 156 | -40.09 (22.39) | -34.75 (22.55)

24. Secondary Outcome: Change From Baseline in Participant Global Assessment (PtGA) of Disease Activity at Week 13, 26, 39, 52, 65, 78, 104, 130 and 156
Description: PtGA: participant assessed their disease activity using a 100 mm visual analog scale ranging from 0 = very good to 100 = worst. Higher scores indicate worse health status.
Time Frame: Baseline, Week 13, 26, 39, 52, 65, 78, 104, 130, 156
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1281 | 413
millimeter
  Baseline: number analyzed (Participants) | 1073 | 354
  Baseline | 54.69 (24.91) | 56.99 (24.57)
  Change at Week 13: number analyzed (Participants) | 1008 | 332
  Change at Week 13 | -13.55 (27.17) | -17.13 (28.34)
  Change at Week 26: number analyzed (Participants) | 823 | 284
  Change at Week 26 | -17.30 (29.43) | -19.32 (27.37)
  Change at Week 39: number analyzed (Participants) | 720 | 230
  Change at Week 39 | -18.09 (28.13) | -21.58 (28.74)
  Change at Week 52: number analyzed (Participants) | 646 | 218
  Change at Week 52 | -19.38 (28.84) | -22.55 (30.03)
  Change at Week 65: number analyzed (Participants) | 566 | 190
  Change at Week 65 | -22.52 (29.15) | -22.74 (28.75)
  Change at Week 78: number analyzed (Participants) | 549 | 180
  Change at Week 78 | -22.24 (30.34) | -24.59 (31.73)
  Change at Week 104: number analyzed (Participants) | 220 | 93
  Change at Week 104 | -22.68 (26.87) | -20.59 (31.57)
  Change at Week 130: number analyzed (Participants) | 204 | 86
  Change at Week 130 | -23.75 (27.23) | -23.10 (29.21)
  Change at Week 156: number analyzed (Participants) | 173 | 83
  Change at Week 156 | -26.30 (27.39) | -21.24 (30.14)

25. Secondary Outcome: Number of Participants in Each Level of the 5 Dimensions of Health Questionnaire by the EuroQol Group (EQ-5D)
Description: EQ-5D: participant rated questionnaire to assess generic health status in two parts: single utility score and visual analog scale. For utility score, participants rated their current health state on 5 dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression with each dimension having three levels of function: 1 indicates no problem; 2 indicates some problem; 3 indicates extreme problem.
Time Frame: Baseline, Week 13, 26, 39, 52, 65, 78, 104, 130, 156
Population: Full analysis set included all participants who received at least 1 dose of Etanercept and had at least 1 effectiveness measurement after start of treatment. Here, "Number Analyzed" signifies number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1281 | 413
Participants
  Baseline: Mobility: number analyzed (Participants) | 1273 | 411
  Baseline: Mobility: No problems | 546 | 177
  Baseline: Mobility: Some problems | 714 | 230
  Baseline: Mobility: Extreme problems | 3 | 0
  Baseline: Mobility: No data | 10 | 4
  Baseline: Self-care: number analyzed (Participants) | 1273 | 411
  Baseline: Self-care: No problems | 798 | 294
  Baseline: Self-care: Some problems | 423 | 107
  Baseline: Self-care: Extreme problems | 37 | 5
  Baseline: Self-care: No data | 15 | 5
  Baseline: Usual Activities: number analyzed (Participants) | 1273 | 411
  Baseline: Usual Activities: No problems | 326 | 115
  Baseline: Usual Activities: Some problems | 887 | 278
  Baseline: Usual Activities: Extreme problems | 51 | 15
  Baseline: Usual Activities: No data | 9 | 3
  Baseline: Pain/Discomfort: number analyzed (Participants) | 1273 | 411
  Baseline: Pain/Discomfort: No problems | 67 | 19
  Baseline: Pain/Discomfort: Some problems | 817 | 264
  Baseline: Pain/Discomfort: Extreme problems | 380 | 125
  Baseline: Pain/Discomfort: No data | 9 | 3
  Baseline: Anxiety/Depression: number analyzed (Participants) | 1273 | 411
  Baseline: Anxiety/Depression: No problems | 693 | 218
  Baseline: Anxiety/Depression: Some problems | 515 | 167
  Baseline: Anxiety/Depression: Extreme problems | 56 | 22
  Baseline: Anxiety/Depression: No data | 9 | 4
  Week 13: Mobility: number analyzed (Participants) | 1240 | 402
  Week 13: Mobility: No problems | 640 | 213
  Week 13: Mobility: Some problems | 586 | 183
  Week 13: Mobility: Extreme problems | 4 | 1
  Week 13: Mobility: No data | 10 | 5
  Week 13: Self-care: number analyzed (Participants) | 1240 | 402
  Week 13: Self-care: No problems | 867 | 304
  Week 13: Self-care: Some problems | 329 | 85
  Week 13: Self-care: Extreme problems | 34 | 7
  Week 13: Self-care: No data | 10 | 6
  Week 13: Usual Activities: number analyzed (Participants) | 1240 | 402
  Week 13: Usual Activities: No problems | 480 | 166
  Week 13: Usual Activities: Some problems | 699 | 222
  Week 13: Usual Activities: Extreme problems | 50 | 10
  Week 13: Usual Activities: No data | 11 | 4
  Week 13: Pain/Discomfort: number analyzed (Participants) | 1240 | 402
  Week 13: Pain/Discomfort: No problems | 162 | 59
  Week 13: Pain/Discomfort: Some problems | 903 | 270
  Week 13: Pain/Discomfort: Extreme problems | 164 | 69
  Week 13: Pain/Discomfort: No data | 11 | 4
  Week 13:Anxiety/ Depression: number analyzed (Participants) | 1240 | 402
  Week 13:Anxiety/ Depression: No problems | 751 | 242
  Week 13:Anxiety/ Depression: Some problems | 427 | 142
  Week 13:Anxiety/ Depression: Extreme problems | 48 | 14
  Week 13:Anxiety/ Depression: No data | 14 | 4
  Week 26: Mobility: number analyzed (Participants) | 1031 | 344
  Week 26: Mobility: No problems | 558 | 200
  Week 26: Mobility: Some problems | 461 | 137
  Week 26: Mobility: Extreme problems | 3 | 0
  Week 26: Mobility: No data | 9 | 7
  Week 26: Self-care: number analyzed (Participants) | 1031 | 344
  Week 26: Self-care: No problems | 733 | 267
  Week 26: Self-care: Some problems | 267 | 66
  Week 26: Self-care: Extreme problems | 22 | 5
  Week 26: Self-care: No data | 9 | 6
  Week 26: Usual Activities: number analyzed (Participants) | 1031 | 344
  Week 26: Usual Activities: No problems | 433 | 156
  Week 26: Usual Activities: Some problems | 550 | 171
  Week 26: Usual Activities: Extreme problems | 38 | 9
  Week 26: Usual Activities: No data | 10 | 8
  Week 26: Pain/Discomfort: number analyzed (Participants) | 1031 | 344
  Week 26: Pain/Discomfort: No problems | 181 | 66
  Week 26: Pain/Discomfort: Some problems | 733 | 234
  Week 26: Pain/Discomfort: Extreme problems | 105 | 36
  Week 26: Pain/Discomfort: No data | 12 | 8
  Week 26: Anxiety/Depression: number analyzed (Participants) | 1031 | 344
  Week 26: Anxiety/Depression: No problems | 641 | 227
  Week 26: Anxiety/Depression: Some problems | 348 | 99
  Week 26: Anxiety/Depression: Extreme problems | 32 | 12
  Week 26: Anxiety/Depression: No data | 10 | 6
  Week 39: Mobility: number analyzed (Participants) | 904 | 279
  Week 39: Mobility: No problems | 506 | 168
  Week 39: Mobility: Some problems | 391 | 108
  Week 39: Mobility: Extreme problems | 3 | 0
  Week 39: Mobility: No data | 4 | 3
  Week 39: Self-care: number analyzed (Participants) | 904 | 279
  Week 39: Self-care: No problems | 664 | 222
  Week 39: Self-care: Some problems | 212 | 49
  Week 39: Self-care: Extreme problems | 21 | 5
  Week 39: Self-care: No data | 7 | 3
  Week 39: Usual Activities: number analyzed (Participants) | 904 | 279
  Week 39: Usual Activities: No problems | 402 | 143
  Week 39: Usual Activities: Some problems | 474 | 131
  Week 39: Usual Activities: Extreme problems | 24 | 3
  Week 39: Usual Activities: No data | 4 | 2
  Week 39: Pain/Discomfort: number analyzed (Participants) | 904 | 279
  Week 39: Pain/Discomfort: No problems | 161 | 67
  Week 39: Pain/Discomfort: Some problems | 641 | 186
  Week 39: Pain/Discomfort: Extreme problems | 98 | 24
  Week 39: Pain/Discomfort: No data | 4 | 2
  Week 39: Anxiety/ Depression: number analyzed (Participants) | 904 | 279
  Week 39: Anxiety/ Depression: No problems | 576 | 183
  Week 39: Anxiety/ Depression: Some problems | 301 | 83
  Week 39: Anxiety/ Depression: Extreme problems | 22 | 11
  Week 39: Anxiety/ Depression: No data | 5 | 2
  Week 52: Mobility: number analyzed (Participants) | 811 | 253
  Week 52: Mobility: No problems | 459 | 158
  Week 52: Mobility: Some problems | 346 | 92
  Week 52: Mobility: Extreme problems | 1 | 0
  Week 52: Mobility: No data | 5 | 3
  Week 52: Self-care: number analyzed (Participants) | 811 | 253
  Week 52: Self-care: No problems | 605 | 210
  Week 52: Self-care: Some problems | 190 | 35
  Week 52: Self-care: Extreme problems | 11 | 5
  Week 52: Self-care: No data | 5 | 3
  Week 52: Usual Activities: number analyzed (Participants) | 811 | 253
  Week 52: Usual Activities: No problems | 400 | 130
  Week 52: Usual Activities: Some problems | 380 | 115
  Week 52: Usual Activities: Extreme problems | 26 | 5
  Week 52: Usual Activities: No data | 5 | 3
  Week 52: Pain/Discomfort: number analyzed (Participants) | 811 | 253
  Week 52: Pain/Discomfort: No problems | 153 | 48
  Week 52: Pain/Discomfort: Some problems | 577 | 185
  Week 52: Pain/Discomfort: Extreme problems | 73 | 17
  Week 52: Pain/Discomfort: No data | 8 | 3
  Week 52: Anxiety/Depression: number analyzed (Participants) | 811 | 253
  Week 52: Anxiety/Depression: No problems | 506 | 168
  Week 52: Anxiety/Depression: Some problems | 268 | 73
  Week 52: Anxiety/Depression: Extreme problems | 28 | 9
  Week 52: Anxiety/Depression: No data | 9 | 3
  Week 65: Mobility: number analyzed (Participants) | 719 | 224
  Week 65: Mobility: No problems | 422 | 141
  Week 65: Mobility: Some problems | 292 | 81
  Week 65: Mobility: Extreme problems | 1 | 0
  Week 65: Mobility: No data | 4 | 2
  Week 65: Self-care: number analyzed (Participants) | 719 | 224
  Week 65: Self-care: No problems | 525 | 183
  Week 65: Self-care: Some problems | 177 | 37
  Week 65: Self-care: Extreme problems | 11 | 2
  Week 65: Self-care: No data | 6 | 2
  Week 65: Usual Activities: number analyzed (Participants) | 719 | 224
  Week 65: Usual Activities: No problems | 361 | 119
  Week 65: Usual Activities: Some problems | 331 | 100
  Week 65: Usual Activities: Extreme problems | 21 | 3
  Week 65: Usual Activities: No data | 6 | 2
  Week 65: Pain/Discomfort: number analyzed (Participants) | 719 | 224
  Week 65: Pain/Discomfort: No problems | 149 | 50
  Week 65: Pain/Discomfort: Some problems | 505 | 147
  Week 65: Pain/Discomfort: Extreme problems | 62 | 23
  Week 65: Pain/Discomfort: No data | 3 | 4
  Week 65: Anxiety/ Depression: number analyzed (Participants) | 719 | 224
  Week 65: Anxiety/ Depression: No problems | 467 | 156
  Week 65: Anxiety/ Depression: Some problems | 225 | 62
  Week 65: Anxiety/ Depression: Extreme problems | 23 | 4
  Week 65: Anxiety/ Depression: No data | 4 | 2
  Week 78: Mobility: number analyzed (Participants) | 692 | 212
  Week 78: Mobility: No problems | 401 | 132
  Week 78: Mobility: Some problems | 286 | 78
  Week 78: Mobility: Extreme problems | 0 | 0
  Week 78: Mobility: No data | 5 | 2
  Week 78: Self-care: number analyzed (Participants) | 692 | 212
  Week 78: Self-care: No problems | 527 | 178
  Week 78: Self-care: Some problems | 155 | 31
  Week 78: Self-care: Extreme problems | 6 | 1
  Week 78: Self-care: No data | 4 | 2
  Week 78: Usual Activities: number analyzed (Participants) | 692 | 212
  Week 78: Usual Activities: No problems | 355 | 115
  Week 78: Usual Activities: Some problems | 316 | 91
  Week 78: Usual Activities: Extreme problems | 16 | 4
  Week 78: Usual Activities: No data | 5 | 2
  Week 78: Pain/Discomfort: number analyzed (Participants) | 692 | 212
  Week 78: Pain/Discomfort: No problems | 152 | 55
  Week 78: Pain/Discomfort: Some problems | 477 | 135
  Week 78: Pain/Discomfort: Extreme problems | 58 | 18
  Week 78: Pain/Discomfort: No data | 5 | 4
  Week 78: Anxiety/Depression: number analyzed (Participants) | 692 | 212
  Week 78: Anxiety/Depression: No problems | 455 | 152
  Week 78: Anxiety/Depression: Some problems | 211 | 50
  Week 78: Anxiety/Depression: Extreme problems | 20 | 7
  Week 78: Anxiety/Depression: No data | 6 | 3
  Week 104: Mobility: number analyzed (Participants) | 278 | 112
  Week 104: Mobility: No problems | 167 | 76
  Week 104: Mobility: Some problems | 109 | 34
  Week 104: Mobility: Extreme problems | 2 | 0
  Week 104: Mobility: No data | 0 | 2
  Week 104: Self-care: number analyzed (Participants) | 278 | 112
  Week 104: Self-care: No problems | 212 | 96
  Week 104: Self-care: Some problems | 61 | 12
  Week 104: Self-care: Extreme problems | 4 | 1
  Week 104: Self-care: No data | 1 | 3
  Week 104: Usual Activities: number analyzed (Participants) | 278 | 112
  Week 104: Usual Activities: No problems | 134 | 68
  Week 104: Usual Activities: Some problems | 141 | 40
  Week 104: Usual Activities: Extreme problems | 3 | 2
  Week 104: Usual Activities: No data | 0 | 2
  Week 104: Pain/Discomfort: number analyzed (Participants) | 278 | 112
  Week 104: Pain/Discomfort: No problems | 48 | 28
  Week 104: Pain/Discomfort: Some problems | 210 | 77
  Week 104: Pain/Discomfort: Extreme problems | 18 | 4
  Week 104: Pain/Discomfort: No data | 2 | 3
  Week 104: Anxiety/ Depression: number analyzed (Participants) | 278 | 112
  Week 104: Anxiety/ Depression: No problems | 190 | 86
  Week 104: Anxiety/ Depression: Some problems | 80 | 21
  Week 104: Anxiety/ Depression: Extreme problems | 8 | 3
  Week 104: Anxiety/ Depression: No data | 0 | 2
  Week 130: Mobility: number analyzed (Participants) | 252 | 107
  Week 130: Mobility: No problems | 144 | 69
  Week 130: Mobility: Some problems | 107 | 38
  Week 130: Mobility: Extreme problems | 0 | 0
  Week 130: Mobility: No data | 1 | 0
  Week 130: Self-care: number analyzed (Participants) | 252 | 107
  Week 130: Self-care: No problems | 188 | 86
  Week 130: Self-care: Some problems | 58 | 20
  Week 130: Self-care: Extreme problems | 4 | 1
  Week 130: Self-care: No data | 2 | 0
  Week 130: Usual Activities: number analyzed (Participants) | 252 | 107
  Week 130: Usual Activities: No problems | 126 | 63
  Week 130: Usual Activities: Some problems | 115 | 43
  Week 130: Usual Activities: Extreme problems | 9 | 1
  Week 130: Usual Activities: No data | 2 | 0
  Week 130: Pain/Discomfort: number analyzed (Participants) | 252 | 107
  Week 130: Pain/Discomfort: No problems | 55 | 30
  Week 130: Pain/Discomfort: Some problems | 174 | 71
  Week 130: Pain/Discomfort: Extreme problems | 22 | 6
  Week 130: Pain/Discomfort: No data | 1 | 0
  Week 130: Anxiety/Depression: number analyzed (Participants) | 252 | 107
  Week 130: Anxiety/Depression: No problems | 176 | 75
  Week 130: Anxiety/Depression: Some problems | 66 | 31
  Week 130: Anxiety/Depression: Extreme problems | 9 | 0
  Week 130: Anxiety/Depression: No data | 1 | 1
  Week 156: Mobility: number analyzed (Participants) | 215 | 95
  Week 156: Mobility: No problems | 126 | 58
  Week 156: Mobility: Some problems | 86 | 35
  Week 156: Mobility: Extreme problems | 2 | 0
  Week 156: Mobility: No data | 1 | 2
  Week 156: Self-care: number analyzed (Participants) | 215 | 95
  Week 156: Self-care: No problems | 156 | 78
  Week 156: Self-care: Some problems | 51 | 12
  Week 156: Self-care: Extreme problems | 7 | 3
  Week 156: Self-care: No data | 1 | 2
  Week 156: Usual Activities: number analyzed (Participants) | 215 | 95
  Week 156: Usual Activities: No problems | 114 | 55
  Week 156: Usual Activities: Some problems | 92 | 35
  Week 156: Usual Activities: Extreme problems | 8 | 3
  Week 156: Usual Activities: No data | 1 | 2
  Week 156: Pain/Discomfort: number analyzed (Participants) | 215 | 95
  Week 156: Pain/Discomfort: No problems | 49 | 21
  Week 156: Pain/Discomfort: Some problems | 149 | 61
  Week 156: Pain/Discomfort: Extreme problems | 15 | 10
  Week 156: Pain/Discomfort: No data | 2 | 3
  Week 156: Anxiety/ Depression: number analyzed (Participants) | 215 | 95
  Week 156: Anxiety/ Depression: No problems | 143 | 68
  Week 156: Anxiety/ Depression: Some problems | 65 | 21
  Week 156: Anxiety/ Depression: Extreme problems | 6 | 4
  Week 156: Anxiety/ Depression: No data | 1 | 2

26. Secondary Outcome: Duration of Morning Stiffness in Participants With Temporary Rigidity
Description: Rigidity was temporary when 'Yes' was given for the question if daily activities could be done without stiffness; rigidity was permanent when 'No' was given for the question if daily activities could be done without stiffness.
Time Frame: Baseline, Week 13, 26, 39, 52, 65, 78, 104, 130, 156
Population: as for outcome 16
Measure: Median (Full Range); unit: Hours
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1281 | 413
Hours
  Baseline: number analyzed (Participants) | 754 | 254
  Baseline | 1.00 [0.0 to 11.0] | 1.00 [0.0 to 11.0]
  Week 13: number analyzed (Participants) | 792 | 264
  Week 13 | 0.50 [0.0 to 10.0] | 0.50 [0.0 to 15.0]
  Week 26: number analyzed (Participants) | 657 | 244
  Week 26 | 0.50 [0.0 to 12.5] | 0.50 [0.0 to 7.0]
  Week 39: number analyzed (Participants) | 606 | 202
  Week 39 | 0.50 [0.0 to 11.7] | 0.50 [0.0 to 7.5]
  Week 52: number analyzed (Participants) | 532 | 183
  Week 52 | 0.50 [0.0 to 10.7] | 0.50 [0.0 to 5.5]
  Week 65: number analyzed (Participants) | 494 | 164
  Week 65 | 0.50 [0.0 to 9.0] | 0.25 [0.0 to 6.0]
  Week 78: number analyzed (Participants) | 480 | 152
  Week 78 | 0.38 [0.0 to 9.0] | 0.46 [0.0 to 10.0]
  Week 104: number analyzed (Participants) | 189 | 91
  Week 104 | 0.25 [0.0 to 8.0] | 0.25 [0.0 to 11.0]
  Week 130: number analyzed (Participants) | 183 | 71
  Week 130 | 0.25 [0.0 to 11.0] | 0.50 [0.0 to 7.0]
  Week 156: number analyzed (Participants) | 157 | 71
  Week 156 | 0.25 [0.0 to 11.0] | 0.33 [0.0 to 4.5]

27. Secondary Outcome: Number of Participants Categorized in Different Classes Depending Upon Percentage of Body Surface Area (BSA) Affected by Psoriatic Arthritis
Description: Participants with psoriatic arthritis were distributed in following different classes depending upon percentage (%) of BSA affected: 1) less than (<) 3 %, 2) 3-10%, 3) 11-20% and 4) >20%. Psoriatic arthritis affecting <3% BSA was considered as mild, 3 to 10 % as moderate and >10 percent as severe.
Time Frame: Baseline, Week 13, 26, 39, 52, 65, 78, 104, 130, 156
Population: Full analysis set. Here, "Number Analyzed" signifies number of participants evaluable for the specified time points. Data for this outcome measure was to be collected and evaluated only for participants with psoriatic arthritis.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 413
Participants
  Baseline: number analyzed (Participants) | 387
  Baseline: <3% | 203
  Baseline: 3-10% | 123
  Baseline: 11-20% | 41
  Baseline: >20% | 20
  Week 13: number analyzed (Participants) | 370
  Week 13: <3% | 247
  Week 13: 3-10% | 82
  Week 13: 11-20% | 28
  Week 13: >20% | 13
  Week 26: number analyzed (Participants) | 316
  Week 26: <3% | 233
  Week 26: 3-10% | 63
  Week 26: 11-20% | 14
  Week 26: >20% | 6
  Week 39: number analyzed (Participants) | 262
  Week 39: <3% | 210
  Week 39: 3-10% | 35
  Week 39: 11-20% | 15
  Week 39: >20% | 2
  Week 52: number analyzed (Participants) | 246
  Week 52: <3% | 196
  Week 52: 3-10% | 37
  Week 52: 11-20% | 10
  Week 52: >20% | 3
  Week 65: number analyzed (Participants) | 215
  Week 65: <3% | 176
  Week 65: 3-10% | 33
  Week 65: 11-20% | 4
  Week 65: >20% | 2
  Week 78: number analyzed (Participants) | 211
  Week 78: <3% | 182
  Week 78: 3-10% | 23
  Week 78: 11-20% | 5
  Week 78: >20% | 1
  Week 104: number analyzed (Participants) | 96
  Week 104: <3% | 80
  Week 104: 3-10% | 12
  Week 104: 11-20% | 2
  Week 104: >20% | 2
  Week 130: number analyzed (Participants) | 89
  Week 130: <3% | 75
  Week 130: 3-10% | 9
  Week 130: 11-20% | 4
  Week 130: >20% | 1
  Week 156: number analyzed (Participants) | 85
  Week 156: <3% | 74
  Week 156: 3-10% | 8
  Week 156: 11-20% | 2
  Week 156: >20% | 1

28. Secondary Outcome: Change From Baseline in Nail Involvement at Week 13, 26, 39, 52, 65, 78, 104, 130 and 156 in Participants With Psoriatic Arthritis
Description: In this outcome measure change in number of nails affected by psoriatic arthritis at specified week compared to baseline is reported. Nails included both finger nails and toe nails.
Time Frame: Baseline, Week 13, 26, 39, 52, 65, 78, 104, 130, 156
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Nails
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 413
Nails
  Baseline: number analyzed (Participants) | 313
  Baseline | 3.18 (4.99)
  Change at Week 13: number analyzed (Participants) | 243
  Change at Week 13 | -0.98 (3.58)
  Change at Week 26: number analyzed (Participants) | 202
  Change at Week 26 | -1.64 (4.38)
  Change at Week 39: number analyzed (Participants) | 167
  Change at Week 39 | -1.75 (4.55)
  Change at Week 52: number analyzed (Participants) | 145
  Change at Week 52 | -2.09 (5.04)
  Change at Week 65: number analyzed (Participants) | 125
  Change at Week 65 | -2.38 (4.89)
  Change at Week 78: number analyzed (Participants) | 126
  Change at Week 78 | -1.79 (4.30)
  Change at Week 104: number analyzed (Participants) | 58
  Change at Week 104 | -1.98 (5.81)
  Change at Week 130: number analyzed (Participants) | 51
  Change at Week 130 | -1.12 (4.75)
  Change at Week 156: number analyzed (Participants) | 53
  Change at Week 156 | -1.38 (5.11)

29. Secondary Outcome: Change From Baseline in Inflamed Dactylitic Digits at Week 13, 26, 39, 52, 65, 78, 104, 130 and 156 in Participants With Psoriatic Arthritis
Description: In this outcome measure change in number of inflamed dactylitic digits at specified week compared to baseline is reported. Dactylitis is inflammation of dactylitic digits (fingers and toes).
Time Frame: Baseline, Week 13, 26, 39, 52, 65, 78, 104, 130, 156
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Dactylitic digits
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 413
Dactylitic digits
  Baseline: number analyzed (Participants) | 309
  Baseline | 0.72 (1.64)
  Change at Week 13: number analyzed (Participants) | 236
  Change at Week 13 | -0.39 (1.36)
  Change at Week 26: number analyzed (Participants) | 195
  Change at Week 26 | -0.54 (1.77)
  Change at Week 39: number analyzed (Participants) | 165
  Change at Week 39 | -0.61 (1.53)
  Change at Week 52: number analyzed (Participants) | 143
  Change at Week 52 | -0.69 (1.58)
  Change at Week 65: number analyzed (Participants) | 121
  Change at Week 65 | -0.50 (2.08)
  Change at Week 78: number analyzed (Participants) | 130
  Change at Week 78 | -0.38 (1.40)
  Change at Week 104: number analyzed (Participants) | 59
  Change at Week 104 | -0.61 (1.47)
  Change at Week 130: number analyzed (Participants) | 57
  Change at Week 130 | -0.63 (1.96)
  Change at Week 156: number analyzed (Participants) | 57
  Change at Week 156 | -0.63 (1.72)

30. Secondary Outcome: Number of Participants With Use of Glucocorticoids and Disease Modifying Antirheumatic Drugs (DMARDs) Baseline Versus Phase 1 (Week 78) and Baseline Versus Phase 2 (Week 156)
Description: In this outcome measure number of participants with use of glucocorticoids and DMARDs at baseline and specified weeks are reported. If participants used glucocorticoids and DMARDs, it was denoted by "Yes" and if they did not use, it was denoted by "No". Data have been reported separately for glucocorticoids and DMARDs at specified weeks respectively, in 4 categories as: 1) Baseline: No and Specified Week: No, 2) Baseline: Yes and Specified Week: No, 3) Baseline: No and Specified Week: Yes, 4) Baseline: Yes and Specified Week: Yes.
Time Frame: Baseline, Week 78, 156
Population: Full analysis set included all participants who received at least 1 dose of Etanercept and had at least 1 effectiveness measurement after start of treatment. Here, "Number Analyzed" = number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1281 | 413
Participants
  Glucocorticoids Usage Baseline Versus Week 78: Baseline: No and Specified Week: No | 499 | 258
  Glucocorticoids Usage Baseline Versus Week 78: Baseline: Yes and Specified Week: No | 177 | 28
  Glucocorticoids Usage Baseline Versus Week 78: Baseline: No and Specified Week: Yes | 312 | 69
  Glucocorticoids Usage Baseline Versus Week 78: Baseline: Yes and Specified Week: Yes | 293 | 58
  DMARDs Usage Baseline Versus Week 78: Baseline: No and Specified Week: No | 124 | 133
  DMARDs Usage Baseline Versus Week 78: Baseline: Yes and Specified Week: No | 655 | 139
  DMARDs Usage Baseline Versus Week 78: Baseline: No and Specified Week: Yes | 24 | 17
  DMARDs Usage Baseline Versus Week 78: Baseline: Yes and Specified Week: Yes | 478 | 124
  Glucocorticoids Usage Baseline Versus Week 156: number analyzed (Participants) | 291 | 116
  Glucocorticoids Usage Baseline Versus Week 156: Baseline: No and Specified Week: No | 168 | 86
  Glucocorticoids Usage Baseline Versus Week 156: Baseline: Yes and Specified Week: No | 91 | 18
  Glucocorticoids Usage Baseline Versus Week 156: Baseline: No and Specified Week: Yes | 20 | 6
  Glucocorticoids Usage Baseline Versus Week 156: Baseline: Yes and Specified Week: Yes | 12 | 6
  DMARDs Usage Baseline Versus Week 156: number analyzed (Participants) | 291 | 116
  DMARDs Usage Baseline Versus Week 156: Baseline: No and Specified Week: No | 33 | 39
  DMARDs Usage Baseline Versus Week 156: Baseline: Yes and Specified Week: No | 234 | 71
  DMARDs Usage Baseline Versus Week 156: Baseline: No and Specified Week: Yes | 1 | 1
  DMARDs Usage Baseline Versus Week 156: Baseline: Yes and Specified Week: Yes | 23 | 5

31. Secondary Outcome: Relationship Between Rheuma Unterstutzungsdienst (RUDI) and Psoriasis Informationsteam (PIT) Participation and Continuation of Treatment With Etanercept
Description: In this outcome number of participants who participated or not participated in RUDI and PIT and impact of their participation in continuation or termination of treatment with Etanercept is reported. For participants whom data was not recorded is reported under category "No Data".
Time Frame: Baseline up to Week 156
Population: Full analysis set included all participants who received at least 1 dose of Etanercept and had at least 1 effectiveness measurement after start of treatment. Here, "Overall Number of participants analyzed" = number of participants evaluable for this measure and "Number Analyzed" = number of participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1241 | 400
Participants
  Rudi and PIT= Yes: number analyzed (Participants) | 347 | 106
  Rudi and PIT= Yes: Treatment Continued | 207 | 58
  Rudi and PIT= Yes: Treatment Terminated | 139 | 48
  Rudi and PIT= Yes: No Data | 1 | 0
  Rudi and PIT= No: number analyzed (Participants) | 894 | 294
  Rudi and PIT= No: Treatment Continued | 555 | 178
  Rudi and PIT= No: Treatment Terminated | 335 | 116
  Rudi and PIT= No: No Data | 4 | 0

32. Secondary Outcome: Relationship Between Rheuma Unterstutzungsdienst (RUDI) and Psoriasis Informationsteam (PIT) Participation and Quality of Life Parameters Using Health Questionnaire by the EuroQol Group (EQ-5D)
Description: In this outcome number of participants who participated or not participated in RUDI and PIT and impact of their participation in quality of life parameters using EQ-5D health questionnaire is reported. For participants whom data was not recorded is reported under category "No Data". EQ-5D: participant rated questionnaire to assess generic health status in two parts: single utility score and visual analog scale. For utility score, participants rated their current health state on 5 dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression with each dimension having three levels of function: 1 indicates no problem; 2 indicates some problem; 3 indicates extreme problem.
Time Frame: Baseline up to Week 156
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 1232 | 398
Participants
  Rudi and PIT= Yes: Mobility: number analyzed (Participants) | 345 | 106
  Rudi and PIT= Yes: Mobility: No problems | 143 | 50
  Rudi and PIT= Yes: Mobility: Some problems | 191 | 54
  Rudi and PIT= Yes: Mobility: Extreme problem | 2 | 0
  Rudi and PIT= Yes: Mobility: No data | 9 | 2
  Rudi and PIT= No: Mobility: number analyzed (Participants) | 887 | 292
  Rudi and PIT= No: Mobility: No problems | 483 | 167
  Rudi and PIT= No: Mobility: Some problems | 394 | 117
  Rudi and PIT= No: Mobility: Extreme problem | 1 | 0
  Rudi and PIT= No: Mobility: No data | 9 | 8
  Rudi and PIT= Yes: Self-care: number analyzed (Participants) | 345 | 106
  Rudi and PIT= Yes: Self-care: No problems | 213 | 72
  Rudi and PIT= Yes: Self-care: Some problems | 111 | 25
  Rudi and PIT= Yes: Self-care: Extreme problem | 13 | 6
  Rudi and PIT= Yes: Self-care: No data | 8 | 3
  Rudi and PIT= No: Self-care: number analyzed (Participants) | 887 | 292
  Rudi and PIT= No: Self-care: No problems | 618 | 233
  Rudi and PIT= No: Self-care: Some problems | 244 | 47
  Rudi and PIT= No: Self-care: Extreme problem | 16 | 4
  Rudi and PIT= No: Self-care: No data | 9 | 8
  Rudi and PIT= Yes: Usual Activities: number analyzed (Participants) | 345 | 106
  Rudi and PIT= Yes: Usual Activities: No problems | 113 | 39
  Rudi and PIT= Yes: Usual Activities: Some problems | 204 | 58
  Rudi and PIT= Yes: Usual Activities: Extreme problem | 19 | 8
  Rudi and PIT= Yes: Usual Activities: No data | 9 | 1
  Rudi and PIT= No: Usual Activities: number analyzed (Participants) | 887 | 292
  Rudi and PIT= No: Usual Activities: No problems | 392 | 142
  Rudi and PIT= No: Usual Activities: Some problems | 456 | 136
  Rudi and PIT= No: Usual Activities: Extreme problem | 30 | 6
  Rudi and PIT= No: Usual Activities: No data | 9 | 8
  Rudi and PIT= Yes: Pain/Discomfort: number analyzed (Participants) | 345 | 106
  Rudi and PIT= Yes: Pain/Discomfort: No problems | 38 | 17
  Rudi and PIT= Yes: Pain/Discomfort: Some problems | 230 | 62
  Rudi and PIT= Yes: Pain/Discomfort: Extreme problem | 68 | 25
  Rudi and PIT= Yes: Pain/Discomfort: No data | 9 | 2
  Rudi and PIT= No: Pain/Discomfort: number analyzed (Participants) | 887 | 292
  Rudi and PIT= No: Pain/Discomfort: No problems | 155 | 60
  Rudi and PIT= No: Pain/Discomfort: Some problems | 611 | 189
  Rudi and PIT= No: Pain/Discomfort: Extreme problem | 112 | 35
  Rudi and PIT= No: Pain/Discomfort: No data | 9 | 8
  Rudi and PIT= Yes: Anxiety/Depression: number analyzed (Participants) | 345 | 106
  Rudi and PIT= Yes: Anxiety/Depression: No problems | 188 | 63
  Rudi and PIT= Yes: Anxiety/Depression: Some problems | 138 | 34
  Rudi and PIT= Yes: Anxiety/Depression: Extreme problem | 11 | 6
  Rudi and PIT= Yes: Anxiety/Depression: No data | 8 | 3
  Rudi and PIT= No: Anxiety/Depression: number analyzed (Participants) | 887 | 292
  Rudi and PIT= No: Anxiety/Depression: No problems | 544 | 188
  Rudi and PIT= No: Anxiety/Depression: Some problems | 300 | 88
  Rudi and PIT= No: Anxiety/Depression: Extreme problem | 34 | 8
  Rudi and PIT= No: Anxiety/Depression: No data | 9 | 8

33. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Treatment-Emergent Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline up to Week 156
Population: Safety analysis set included all patients who received at least 1 dose of Etanercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Unclear Diagnosis
Number analyzed (Participants) | 1378 | 440 | 3
Participants
  AEs | 658 | 190 | 1
  SAEs | 159 | 47 | 0

34. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) by Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious adverse events. AEs were classified according to the severity in 3 categories a)mild: AEs not interfered with participant's usual function b)moderate: AEs interfered to some extent with participant's usual function c)severe: AEs interfered significantly with participant's usual function. Participants may be counted in more than 1 category.
Time Frame: Baseline up to Week 156
Population: Safety analysis set included all patients who received at least 1 dose of Etanercept. Here, "Overall Number of Participants Analyzed" signifies number of participants who had at least 1 treatment AE.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Unclear Diagnosis
Number analyzed (Participants) | 658 | 190 | 1
Participants
  Mild | 292 | 85 | 0
  Moderate | 377 | 104 | 0
  Severe | 172 | 52 | 0
  No Data | 36 | 7 | 1

35. Other Pre Specified Outcome: Number of Participants With Discontinuation of Etanercept Treatment
Description: Number of participants those who discontinued Etanercept treatment at Week 78 and 156 are reported in this outcome measure.
Time Frame: Week 78, 156
Population: Safety analysis set included all patients who received at least 1 dose of Etanercept. Here, "Number Analyzed" signifies number of participants evaluable for specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Unclear Diagnosis
Number analyzed (Participants) | 1378 | 440 | 3
Participants
  Week 78 | 57 | 18 | 1
  Week 156: number analyzed (Participants) | 291 | 116 | 0
  Week 156 | 8 | 4 |

36. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Treatment Related Adverse Events
Description: Treatment-related AE was any untoward medical occurrence in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious adverse events. Relatedness to study treatment was assessed by the investigator.
Time Frame: Baseline up to Week 156
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Unclear Diagnosis
Number analyzed (Participants) | 658 | 190 | 1
Participants | 345 | 100 | 1

37. Other Pre Specified Outcome: Number of Participants With Results of Tolerability Assessment by Physician and Participant
Description: Physicians and participants rated the tolerability of Etanercept treatment by means of a 4-point scale as: 1) very good, 2) good, 3) moderate and 4) insufficient.
Time Frame: Week 78, 156
Population: Safety analysis set included all patients who received at least 1 dose of Etanercept. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Unclear Diagnosis
Number analyzed (Participants) | 1378 | 440 | 3
Participants
  Week 78: Physician Assessment: number analyzed (Participants) | 699 | 220 | 1
  Week 78: Physician Assessment: Very good | 439 | 146 | 1
  Week 78: Physician Assessment: Good | 252 | 70 | 0
  Week 78: Physician Assessment: Moderate | 4 | 2 | 0
  Week 78: Physician Assessment: Insufficient | 4 | 2 | 0
  Week 78: Participant Assessment: number analyzed (Participants) | 607 | 183 | 1
  Week 78: Participant Assessment: Very good | 284 | 96 | 1
  Week 78: Participant Assessment: Good | 281 | 75 | 0
  Week 78: Participant Assessment: Moderate | 33 | 12 | 0
  Week 78: Participant Assessment: Insufficient | 9 | 0 | 0
  Week 156: Physician Assessment: number analyzed (Participants) | 220 | 97 | 0
  Week 156: Physician Assessment: Very good | 149 | 67 |
  Week 156: Physician Assessment: Good | 70 | 30 |
  Week 156: Physician Assessment: Moderate | 1 | 0 |
  Week 156: Physician Assessment: Insufficient | 0 | 0 |
  Week 156: Participant Assessment: number analyzed (Participants) | 210 | 94 | 0
  Week 156: Participant Assessment: Very good | 115 | 55 |
  Week 156: Participant Assessment: Good | 89 | 38 |
  Week 156: Participant Assessment: Moderate | 4 | 1 |
  Week 156: Participant Assessment: Insufficient | 2 | 0 |

38. Other Pre Specified Outcome: Number of Participants With Pregnancy, Puerperium and Perinatal Conditions
Description: In this outcome measure total number of participants with pregnancy, puerperium and perinatal conditions are reported. Pregnancy, puerperium and perinatal conditions included pregnancy, abortion, abortion spontaneous or premature baby.
Time Frame: Baseline up to Week 156
Population: Safety analysis set included all patients who received at least 1 dose of Etanercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Unclear Diagnosis
Number analyzed (Participants) | 1378 | 440 | 3
Participants | 4 | 1 | 0

39. Other Pre Specified Outcome: Number of Participants Who Used Concomitant Medication
Description: Number of participants who used medication other than Etanercept for relief of pain. It was determined by the treating physician.
Time Frame: Baseline up to Week 156
Population: Safety analysis set included all patients who received at least 1 dose of Etanercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Unclear Diagnosis
Number analyzed (Participants) | 1378 | 440 | 3
Participants | 1284 | 376 | 2

ADVERSE EVENTS:
Time Frame: Baseline up to Week 156
Description: Same event may appear both an AE and SAE. However, what is presented are distinct events. Event may be serious in 1 and nonserious in other participant or 1 participant may have experienced both serious and nonserious AE.
Arm/Group | Participants With Rheumatoid Arthritis | Participants With Psoriatic Arthritis | Participants With Unclear Diagnosis
All-Cause Mortality (participants affected / at risk) | 6/1378 | 0/440 | 0/3
Serious Adverse Events (participants affected / at risk) | 159/1378 | 47/440 | 0/3
Other Adverse Events (participants affected / at risk) | 579/1378 | 167/440 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Rheumatoid Arthritis (N=1378) | Participants With Psoriatic Arthritis (N=440) | Participants With Unclear Diagnosis (N=3)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 4 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 3 | 0
Coronary artery disease (Cardiac disorders) | 4 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 2 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Trisomy 8 (Congenital, familial and genetic disorders) | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 2 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Macular hole (Eye disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Condition aggravated (General disorders) | 7 | 3 | 0
Disease progression (General disorders) | 2 | 1 | 0
Injection site pruritus (General disorders) | 2 | 0 | 0
Pain (General disorders) | 1 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0
Disease recurrence (General disorders) | 1 | 0 | 0
Drug ineffective (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0
Medical device complication (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0
Necrosis (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 0
Abscess (Infections and infestations) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 0
Osteomyelitis (Infections and infestations) | 2 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0
Staphylococcal infection (Infections and infestations) | 2 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 1 | 0
Abscess oral (Infections and infestations) | 1 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1 | 0
Arteriosclerotic gangrene (Infections and infestations) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Bursitis infective (Infections and infestations) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Sinusitis aspergillus (Infections and infestations) | 1 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Impacted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Venous injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood pressure abnormal (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 6 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Loose body in joint (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chest wall tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Warty dyskeratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 0
Facial paresis (Nervous system disorders) | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 1 | 0
Borderline mental impairment (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 3 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Clinically isolated syndrome (Nervous system disorders) | 0 | 1 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 0 | 0
Meralgia paraesthetica (Nervous system disorders) | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Neuritis (Nervous system disorders) | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0
Vascular encephalopathy (Nervous system disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 0
Nephritis (Renal and urinary disorders) | 1 | 0 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 2 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary vein occlusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arthrodesis (Surgical and medical procedures) | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Rheumatoid Arthritis (N=1378) | Participants With Psoriatic Arthritis (N=440) | Participants With Unclear Diagnosis (N=3)
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 3 | 0 | 0
Palpitations (Cardiac disorders) | 3 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Cyanosis (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 10 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 4 | 0 | 0
Eye irritation (Eye disorders) | 2 | 1 | 0
Scleritis (Eye disorders) | 2 | 1 | 0
Dry eye (Eye disorders) | 1 | 1 | 0
Uveitis (Eye disorders) | 1 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Chalazion (Eye disorders) | 1 | 0 | 0
Corneal disorder (Eye disorders) | 1 | 0 | 0
Episcleritis (Eye disorders) | 1 | 0 | 0
Erythema of eyelid (Eye disorders) | 1 | 0 | 0
Eye inflammation (Eye disorders) | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 2 | 0 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Iridocyclitis (Eye disorders) | 1 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0
Macular degeneration (Eye disorders) | 1 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 4 | 2 | 0
Hypersensitivity (Immune system disorders) | 4 | 2 | 0
Seasonal allergy (Immune system disorders) | 1 | 1 | 0
Atopy (Immune system disorders) | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 6 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 | 1 | 0
Haematuria (Renal and urinary disorders) | 3 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0
Menstrual discomfort (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 23 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 11 | 5 | 0
Dry mouth (Gastrointestinal disorders) | 5 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0
Gastritis (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 0
Gingival ulceration (Gastrointestinal disorders) | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Drug ineffective (General disorders) | 60 | 24 | 0
Injection site reaction (General disorders) | 55 | 10 | 0
Injection site erythema (General disorders) | 22 | 5 | 1
Injection site pruritus (General disorders) | 14 | 4 | 0
Injection site hypersensitivity (General disorders) | 14 | 2 | 0
Fatigue (General disorders) | 10 | 4 | 0
Pyrexia (General disorders) | 9 | 4 | 0
Oedema peripheral (General disorders) | 8 | 4 | 0
Condition aggravated (General disorders) | 6 | 1 | 0
Chest pain (General disorders) | 2 | 3 | 0
Pain (General disorders) | 5 | 0 | 0
Chills (General disorders) | 3 | 1 | 0
Injection site pain (General disorders) | 2 | 2 | 0
Injection site swelling (General disorders) | 4 | 0 | 0
Local swelling (General disorders) | 1 | 3 | 0
Cyst (General disorders) | 1 | 2 | 0
Injection site dermatitis (General disorders) | 2 | 1 | 0
Injection site rash (General disorders) | 3 | 0 | 0
Injection site urticaria (General disorders) | 3 | 0 | 0
Swelling (General disorders) | 2 | 1 | 0
Asthenia (General disorders) | 2 | 0 | 0
Feeling abnormal (General disorders) | 1 | 1 | 0
Impaired healing (General disorders) | 1 | 1 | 0
Injection site discomfort (General disorders) | 1 | 1 | 0
Local reaction (General disorders) | 2 | 0 | 0
Oedema (General disorders) | 2 | 0 | 0
Administration site reaction (General disorders) | 1 | 0 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0
Feeling cold (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Injection site irritation (General disorders) | 1 | 0 | 0
Injection site vesicles (General disorders) | 1 | 0 | 0
Instillation site reaction (General disorders) | 1 | 0 | 0
Mucosal dryness (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0
Performance status decreased (General disorders) | 1 | 0 | 0
Influenza (Infections and infestations) | 42 | 16 | 0
Respiratory tract infection (Infections and infestations) | 23 | 8 | 0
Bronchitis (Infections and infestations) | 17 | 9 | 0
Nasopharyngitis (Infections and infestations) | 18 | 6 | 0
Herpes zoster (Infections and infestations) | 17 | 1 | 0
Infection (Infections and infestations) | 11 | 4 | 0
Sinusitis (Infections and infestations) | 9 | 5 | 0
Urinary tract infection (Infections and infestations) | 12 | 2 | 0
Cystitis (Infections and infestations) | 10 | 0 | 0
Rhinitis (Infections and infestations) | 5 | 3 | 0
Conjunctivitis (Infections and infestations) | 6 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 2 | 0
Herpes simplex (Infections and infestations) | 5 | 1 | 0
Laryngitis (Infections and infestations) | 3 | 3 | 0
Pneumonia (Infections and infestations) | 6 | 0 | 0
Bronchopneumonia (Infections and infestations) | 2 | 2 | 0
Otitis media (Infections and infestations) | 3 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 20 | 4 | 0
Oral herpes (Infections and infestations) | 6 | 2 | 0
Tooth infection (Infections and infestations) | 2 | 2 | 0
Erysipelas (Infections and infestations) | 2 | 1 | 0
Erythema migrans (Infections and infestations) | 3 | 0 | 0
Fungal infection (Infections and infestations) | 3 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 2 | 1 | 0
Pulpitis dental (Infections and infestations) | 3 | 0 | 0
Rash pustular (Infections and infestations) | 2 | 1 | 0
Viral infection (Infections and infestations) | 2 | 1 | 0
Abscess (Infections and infestations) | 1 | 1 | 0
Acute tonsillitis (Infections and infestations) | 2 | 0 | 0
Furuncle (Infections and infestations) | 1 | 1 | 0
Gastrointestinal viral infection (Infections and infestations) | 2 | 0 | 0
Herpes virus infection (Infections and infestations) | 2 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 1 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0
Abscess oral (Infections and infestations) | 1 | 0 | 0
Adenoviral hepatitis (Infections and infestations) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Borrelia infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0
Dental fistula (Infections and infestations) | 0 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0
Gastric infection (Infections and infestations) | 1 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1 | 0
Infection susceptibility increased (Infections and infestations) | 1 | 0 | 0
Latent tuberculosis (Infections and infestations) | 1 | 0 | 0
Mastoiditis (Infections and infestations) | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0
Oral infection (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 3 | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 3 | 0
Wound (Injury, poisoning and procedural complications) | 4 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pneumoconiosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 5 | 3 | 0
Liver function test abnormal (Investigations) | 6 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 5 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 2 | 0
Weight decreased (Investigations) | 5 | 0 | 0
Hepatic enzyme increased (Investigations) | 2 | 2 | 0
Transaminases increased (Investigations) | 2 | 2 | 0
Arthroscopy (Investigations) | 2 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 0
Weight increased (Investigations) | 2 | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Biopsy liver (Investigations) | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0
Blood pressure abnormal (Investigations) | 1 | 0 | 0
Bone scan abnormal (Investigations) | 0 | 1 | 0
C-reactive protein (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase abnormal (Investigations) | 1 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 0
Lymphoblast morphology abnormal (Investigations) | 1 | 0 | 0
Radioisotope scan (Investigations) | 1 | 0 | 0
Respiratory rate increased (Investigations) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 13 | 4 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Dactylitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Rheumatic fever (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Headache (Nervous system disorders) | 12 | 2 | 0
Restless legs syndrome (Nervous system disorders) | 5 | 0 | 0
Sciatica (Nervous system disorders) | 3 | 2 | 0
Hypertonia (Nervous system disorders) | 1 | 2 | 0
Cervicobrachial syndrome (Nervous system disorders) | 2 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 0
Memory impairment (Nervous system disorders) | 2 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Morton's neuralgia (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 9 | 6 | 0
Restlessness (Psychiatric disorders) | 4 | 1 | 0
Sleep disorder (Psychiatric disorders) | 3 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Emotional distress (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0
Listless (Psychiatric disorders) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 13 | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 9 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 6 | 0
Eczema (Skin and subcutaneous tissue disorders) | 5 | 3 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 6 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Leukoplakia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cataract operation (Surgical and medical procedures) | 4 | 0 | 0
Dental operation (Surgical and medical procedures) | 0 | 4 | 0
Joint injection (Surgical and medical procedures) | 2 | 0 | 0
Surgery (Surgical and medical procedures) | 2 | 0 | 0
Synovectomy (Surgical and medical procedures) | 2 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 2 | 0 | 0
Wound treatment (Surgical and medical procedures) | 2 | 0 | 0
Bunion operation (Surgical and medical procedures) | 1 | 0 | 0
Carpal tunnel decompression (Surgical and medical procedures) | 1 | 0 | 0
Cyst removal (Surgical and medical procedures) | 1 | 0 | 0
Dental implantation (Surgical and medical procedures) | 1 | 0 | 0
Elbow operation (Surgical and medical procedures) | 1 | 0 | 0
Endodontic procedure (Surgical and medical procedures) | 0 | 1 | 0
Glaucoma surgery (Surgical and medical procedures) | 0 | 1 | 0
Hernia repair (Surgical and medical procedures) | 1 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0 | 0
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0 | 0
Joint surgery (Surgical and medical procedures) | 0 | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 0
Lens extraction (Surgical and medical procedures) | 1 | 0 | 0
Polypectomy (Surgical and medical procedures) | 1 | 0 | 0
Rehabilitation therapy (Surgical and medical procedures) | 0 | 1 | 0
Removal of internal fixation (Surgical and medical procedures) | 1 | 0 | 0
Rheumatoid nodule removal (Surgical and medical procedures) | 0 | 1 | 0
Skin neoplasm excision (Surgical and medical procedures) | 1 | 0 | 0
Synoviorthesis (Surgical and medical procedures) | 1 | 0 | 0
Tendon operation (Surgical and medical procedures) | 0 | 1 | 0
Tonsillectomy (Surgical and medical procedures) | 1 | 0 | 0
Wisdom teeth removal (Surgical and medical procedures) | 1 | 0 | 0
Hypertension (Vascular disorders) | 5 | 3 | 0
Thrombosis (Vascular disorders) | 3 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Haematoma (Vascular disorders) | 2 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 0 | 0
Venous thrombosis (Vascular disorders) | 2 | 0 | 0
Arterial stenosis (Vascular disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Intra-abdominal haematoma (Vascular disorders) | 1 | 0 | 0
Labile hypertension (Vascular disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 5 | 0 | 0
Enteritis (Gastrointestinal disorders) | 3 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Lumbar hernia (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 1 | 0
Tooth loss (Gastrointestinal disorders) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 1 | 0
Bursitis infective (Infections and infestations) | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Essential hypertension (Vascular disorders) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-09-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT01623752/Prot_SAP_000.pdf